CLINICAL TRIAL: NCT00166140
Title: Heparin Responses in Pediatric Patients Undergoing Cardiopulmonary Bypass.
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nina Guzzetta, M.D., Assistant Professor of Anesthesiology, Emory University
Other Study IDs: 549-2002
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Children With Heart Defects
Keywords: pediatrics; cardiac; surgery

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Heparin is an anticoagulant or "blood thinner". Heparin is always given to patients undergoing open-heart surgery to prevent blood from clotting when a patient is placed on the heart-lung machine. Heparin works by combining with a protein in blood to prevent other proteins from working together to form a clot. The protein that heparin combines with seems to be different in infants and young children compared to adults.

The purpose of this study is to determine which proteins in children have a direct impact on the way heparin works. We also want to see how this may change at different ages. We will enroll two age groups of children; birth to 2 years and 10 years or older. A total of 125 patients will be enrolled into this study. These patients will already be scheduled for open-heart surgery using a heart-lung machine.

The testing involves taking blood samples when the patient is asleep for surgery; and later from their intravenous line, IV. They will all have IV's in place already because of the surgery. Therefore the study will cause no pain or discomfort for the patients who take part.

DETAILED DESCRIPTION:
Introduction

Anticoagulation during cardiopulmonary bypass (CPB) is necessary to prevent clotting as blood comes in contact with the unphysiologic surfaces of the extracorporeal circuit, and is achieved by administration of unfractionated heparin which binds to antithrombin III (ATIII) to potentiate and accelerate its inhibition of thrombin and other activated coagulation factors. In adults, heparin dose responses are decreased as ATIII concentrations fall. Findings in adults indicate that the administration of supplemental ATIII as concentrations fall below 80 u/dl may help to preserve heparin's effectiveness during CPB(1). Since ATIII levels in infants do not reach 80 u/dl until 3-6 months of age (2), one would likewise anticipate that heparin dose-response relationships would be affected. However, preliminary investigations in children less than one year of age show that there is no correlation between preoperative ATIII concentrations with the projected heparin dose-response (HDR) curve or with changes in the activated clotting time (ACT) value after heparin administration(3). The lack of correlation of ATIII levels with these heparin dose responses in infants raises important questions for pediatric patients regarding the mechanism by which heparin exerts its anticoagulant effects as well as the adequacy of heparinization during CPB.

Another coagulation inhibitor, heparin cofactor II (HCII), forms a stable enzyme-inhibitor complex that inhibits thrombin in a reaction enhanced by heparin(4). Although in the adult population, the exact role of HCII is unclear, perhaps in neonates its role is more significant. Alpha-2-macroglobulin (2M), a less important inhibitor of thrombin in adults, has concentrations well above adult values in newborns and continues to increase in concentration during the first 6 months of life(2). In neonates, 2M has been shown to have an important role as a thrombin inhibitor although its association with heparin responses during CPB is unknown.

The adequacy of anticoagulation during CPB can be assessed by the extent to which heparin attenuates the formation and activation of thrombin. However, the very short half-life of thrombin in the presence of heparin and ATIII prohibits the direct measurement of thrombin concentration while on CPB. The peptide prothrombin fragment 1.2 (PT1.2), which is formed as prothrombin is converted to thrombin, is readily measurable and provides a way of evaluating thrombin formation during CPB(5). One of thrombin's major actions, the conversion of fibrinogen to fibrin, releases another measurable peptide, fibrinopeptide A (FPA), thereby providing a means of assessing thrombin activity during CPB(5).

In an attempt to determine the mechanism by which heparin exerts its anticoagulant effect in children, this investigation proposes to evaluate the relationship between preoperative ATIII, HCII and 2M levels in pediatric patients of varying age groups with clinical measurements of heparin response in the operating room, specifically changes in ACT values with heparin administration and a generated heparin dose-response curve. We also propose to evaluate the adequacy of heparinization in neonates, whom are known to have a quantitative deficiency in ATIII, by measuring PT1.2 and FPA that is produced during CPB as compared to an adult population.

Background The management of the coagulation system during pediatric cardiac surgery is a complex task. Cardiopulmonary bypass is a significant thrombogenic stimulus requiring anticoagulation with heparin prior to its initiation, and after the completion of the bypass period, reversal of heparin and the reestablishment of hemostasis prior to surgical closure. These manipulations toward both hypo- and hypercoagulability must be accomplished during the care of these children. The inability to attain either of these states within precise limits at specified points during the surgical procedure can have far-reaching implications. Adequate inhibition of the coagulation cascades is obviously necessary during CPB to prevent catastrophic clot formation in the CPB circuit. A state of partial, but inadequate, anticoagulation during this time can still prevent clot formation but will lead to the formation of coagulation products that can have deleterious effects on coagulation after CPB: thrombin is generated and subsequently activates plasminogen and the fibrinolytic system; fibrinolysis prevents the reestablishment of hemostasis and perpetuates the activation of the coagulation system; and thrombin, plasmin, and fibrin degradation products all severely disrupt post-CPB platelet function.

Anticoagulation during CPB is accomplished by the administration of heparin, which is empirically dosed on the basis of patient weight. The degree of heparin-induced anticoagulation during cardiac surgery can be measured in the operating room by assessing heparin levels or by assessing heparin's anticoagulant effect with activated clotting times (ACTs). The most commonly used method is ACT monitoring. Unfortunately, the ACT is influenced by factors other than heparin, such as hemodilution and hypothermia. While not of major concern in adults and older children, the hemodilution accompanying CPB is extreme in neonates and young infants. Similarly, while most adult cardiac surgery is performed under normothermic or mild hypothermic conditions, the surgical procedures in infants are often conducted at extremely hypothermic temperatures. Therefore, ACT measurements during cardiac surgery in infants may not be reflective of the degree of heparin-induced anticoagulation. Indeed, heparin levels in young children are significantly lower than those found, maintained, and considered safe during CPB in adults while the ACT measurements in these children remain in the range felt to indicate adequate anticoagulation (6,7)

In full term and preterm infants the coagulation system begins to develop gradually during gestation and continues to mature toward the adult system during the postnatal period. By 6 months of age, most components of the coagulation system, both procoagulants and inhibitors, are well within the normal adult range(8). However, at birth the coagulation system is quantitatively immature with significant deficiencies in many factor levels. One of these deficient factors is AT III. AT III levels are only 60% of adult values at birth and do not attain adult levels until 3 to 6 months of age. In the face of these low AT III levels, the ability of heparin to produce adequate anticoagulation during cardiac surgery in infants becomes a significant concern, and it is reasonable to consider that there are potential differences in coagulation between neonates and adults undergoing CPB. Questions arise as to the role that diminished AT III levels have in producing an anticoagulant effect in young infants. Further questions arise as to the adequacy of anticoagulation during cardiac surgery in young infants since, the accepted standard of care, only ACT measurements, are routinely used to make this determination. The first question can be addressed by the comparison of AT III levels as well as other potential heparin cofactor levels with more specific indicators of the inhibition of the coagulation system. The second question can be addressed by the measurement of specific breakdown products released during the formation of thrombin upon activation of the coagulation system.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective cardiac surgery requiring the use of cardiopulmonary bypass scheduled at Children's Healthcare of Atlanta, Egleston (either a first procedure or a reoperation)
2. Patients within the appropriate age groups (birth to 2 years of age, and 10 years or older)
3. Parents or legal guardian willing for child to participate and able to sign the provided informed consent -

Exclusion Criteria:

1. Patients undergoing cardiac surgery not requiring the use of CPB
2. Patients undergoing any emergent procedure/surgery
3. Patients who take preoperative anticoagulant therapy
4. Patients with a CPB time greater that 4 hours
5. Patients requiring a return to CPB for any reason
6. Patients whose parents or legal guardian are unwilling or unable to sign the provided informed consent
7. Patients who, in the opinion of the investigators, should not be included in the study
8. Patients who are older than 2 years, but less than 10 years of age are excluded

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing elective cardiac surgery requiring the use of cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 125
Dates: Start 2002-12; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina A Guzzetta, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States

REFERENCES:
- [Background] Despotis GJ, Levine V, Joist JH, Joiner-Maier D, Spitznagel E. Antithrombin III during cardiac surgery: effect on response of activated clotting time to heparin and relationship to markers of hemostatic activation. Anesth Analg. 1997 Sep;85(3):498-506. doi: 10.1097/00000539-199709000-00005. PMID 9296400
- [Background] Andrew M, Paes B, Johnston M. Development of the hemostatic system in the neonate and young infant. Am J Pediatr Hematol Oncol. 1990 Spring;12(1):95-104. doi: 10.1097/00043426-199021000-00019. PMID 2178462
- [Background] Horkay F, Martin P, Rajah SM, Walker DR. Response to heparinization in adults and children undergoing cardiac operations. Ann Thorac Surg. 1992 May;53(5):822-6. doi: 10.1016/0003-4975(92)91444-e. PMID 1570978
- [Background] McIntosh MA, Earhart CF. Coordinate regulation by iron of the synthesis of phenolate compounds and three outer membrane proteins in Escherichia coli. J Bacteriol. 1977 Jul;131(1):331-9. doi: 10.1128/jb.131.1.331-339.1977. PMID 141448